CLINICAL TRIAL: NCT05187416
Title: Correlation Between Elastic Modulus of Ultrasonic Shear Wave and Tumor Stromal Component in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20212175-C-1
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Neoplasms
Keywords: 2D-SWE
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: two-dimensional shear wave elastography — Preoperative ultrasound elastography examination

SUMMARY:
Pancreatic cancer is a gastrointestinal tumor with a high degree of malignancy. Currently, there are many first-line chemotherapy regimens in clinical practice, but the individual selection of chemotherapy regimens has not been unanimously recognized.This study is aimed at exploring the correlation between the two-dimensional shear wave elastography (2D - SWE) parameters and pancreatic cancer stromal elements proportion through an ultrasound scan for resectable pancreatic cancer cases and postoperative pathological specimen analysis. Then determine if the pancreatic cancer two-dimensional shear wave elastography can guide clinicians selecting chemotherapy scheme by predicting tumor stromal elements .These results are expected to provide an effective non-invasive diagnostic basis for individualized treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria

1. Patients with resectable pancreatic cancer underwent ultrasound examination before surgery
2. Conventional ultrasound can clearly show pancreatic space-occupying lesions and the elastic measurements show good images
3. The patient agrees to receive ultrasound elasticity examination and signs informed consent
4. All patients had no history of radiotherapy or chemotherapy before ultrasound examination
5. All clinical case data and auxiliary examination data are complete and accessible.

Exclusion Criteria

1. Ultrasound evaluation was not performed before ultrasound-guided needle biopsy
2. Conventional ultrasound could not clearly show pancreatic space-occupying lesions or poor elastic measurement images
3. Patients who refuse to accept examination or give up treatment
4. Patients receiving neoadjuvant chemotherapy or radiotherapy before ultrasound examination
5. Incomplete clinical data and auxiliary examination data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cases of pancreatic cancer in Xijing Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Elastic modulus measured by Ultrasonic shear wave and tumor stromal component assessed by pathological analysis in pancreatic cancer | Baseline (Preoperative ultrasound elastography examination)

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No